CLINICAL TRIAL: NCT05973604
Title: Prevalence of Primary Aldosteronism in Patients With Atrial Fibrillation (ERETRIA Trial)
Brief Title: Prevalence of Primary Aldosteronism in Atrial Fibrillation
Acronym: ERETRIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Maria Toumpourleka, Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: 4418/26/01/2021
Record Dates: First submitted 2023-07-19; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation; Primary Aldosteronism
Keywords: Atrial Fibrillation; Primary Aldosteronism
MeSH Terms: conditions — Atrial Fibrillation; Hyperaldosteronism | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Screening and Confirmatory diagnostic test for primary aldosteronism — Screening for primary aldosteronism will be performed with measurement of aldosterone-to-renin ratio after 2 hours of bed rest. Renin measurement will be performed by estimating plasma renin activity. The screening test will be considered positive when the ratio is >30, accompanied by elevated aldosterone values (>15 ng/ml). Patients with a positive result will undergo further confirmatory testing with intravenous sodium test (administration 2 liters of normal saline N/S 0.9%, over a period of 4 hours, while the patient is supine. Considered positive if aldosterone levels are >5mg/dl at the end of the test). Alternative confirmatory methods are captopril test (Administration of 50 mg of captopril. Considered positive when aldosterone levels are >8.5 mg/dl 2 hours after the intake) or hydrocortisone test (Administration of 0.1mg of hydrocortisone 4 times a day for a period of 4 days. Considered positive if elevated aldosterone levels (>6ng/dl) are found at the end of the test).

SUMMARY:
This is an observational prospective cross-sectional study, investigating the prevalence of primary aldosteronism in patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of atrial fibrillation with a standard surface ECG tracing of at least 30 seconds (either paroxysmal or persistent or permanent).

Exclusion Criteria:

* Diagnosis of primary aldosteronism
* Diagnosis of heart failure, treated with mineralocorticoid receptor antagonists
* Inability to be subjected to any confirmatory tests for primary aldosteronism
* Acute vascular event (acute coronary syndrome, stroke, acute peripheral vascular event) within last 6 months
* Renal replacement therapy
* Incompetence of unwillingness to provide written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of primary aldosteronism in patients with atrial fibrillation | Baseline
  Percentage of patients with positive screening and confirmatory test for primary aldosteronism

SECONDARY OUTCOMES:
Association of marker of arterial stiffness with presence of primary aldosteronism in patients with atrial fibrillation | Baseline
  Pulse wave velocity
Association of echocardiographic indices with presence of primary aldosteronism in patients with atrial fibrillation. | Baseline
  Left ventricular global longitudinal strain (GLS) measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Maria Toumpourleka, MSc, Principal Investigator — Third Cardiology Department, Aristotle University of Thessaloniki, Thessaloniki, Greece; Vassilios P Vassilikos, PhD, Study Director — Third Cardiology Department, Aristotle University of Thessaloniki, Thessaloniki, Greece; Michael Doumas, PhD, Study Director — Second Propedeutic Department of Internal Medicine, Aristotle University of Thessaloniki, Thessaloniki, Greece; Christodoulos E Papadoupoulos, Study Chair — Third Cardiology Department, Aristotle University of Thessaloniki, Thessaloniki, Greece
Locations (1):
- Ippokratio General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided